CLINICAL TRIAL: NCT00745329
Title: The Effect of Infliximab,Adalimumab, Azathioprines and 5-Aminosalicylate on Semen Quality in Men With Inflammatory Bowel Disease
Brief Title: The Effect of Infliximab on Sperm Quality
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Dr Sigal Fishman Gastroenterology institution Tel Aviv Sourasky Medical Center, Tel Aviv Sourasky Medical Center
Other Study IDs: TASMC-08-SF-182-CTIL
Record Dates: First submitted 2008-09-01; First posted 2008-09-03 (Estimated); Last update posted 2008-09-03 (Estimated); Status verified 2008-09

CONDITIONS: Crohn's Disease; Ulcerative Colitis
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 2: 1. patients
  2. healthy volunteers
  Interventions: Other: sperm quality test

INTERVENTIONS:
Other: sperm quality test — All participants will undergo sequential sperm quality tests and blood tests

SUMMARY:
Background: The treatment of inflammatory bowel diseases (IBD) is based mainly on 3 compounds: 1- 5 aminosalysilates . 2- immunomodulators (Azathioprines). 3- Biologic therapies (Infliximab, Adalimumab) . There are no established data in the literature whether these therapies effects sperm quality. Given that a large number of the patients are young men in the reproductive stage of their lives , It of importance to investigate these effect.

Aim: To investigate the effect of chronic treatment of any of the three therapy mentioned above, on sperm quality .

ELIGIBILITY:
Inclusion Criteria:

* Male above the age of 18
* Capable of giving informed consent
* Diagnosed with IBD at least 3 months
* Patients that are going to start a treatment with on of the following groups: 5ASA, Azathioprines, infliximab or ADAlimumab
* Patients that are treated with therapies mentioned in article 4 for at least 3 months

Exclusion Criteria:

* Male younger than 18

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with inflammatory bowel disease (IBD) and healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2008-10